CLINICAL TRIAL: NCT04670120
Title: Evaluation of Early Bactericidal Activity and Safety in Pulmonary Tuberculosis With Pyrifazimine (TBI-166)
Brief Title: Early Bactericidal Activity Safety Pulmonary Tuberculosis Pyrifazimine (TBI-166)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Shandong Chest Hospital (Unknown); Zhengzhou Sixth People's Hospital (Unknown)
Responsible Party: Principal Investigator, Chu naihu, TB Director, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB-Pyrifazimine (TBI-166)
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Sensitive Pulmonary Tuberculosis
Keywords: tuberculosis; pyfazimine; early bactericidal activity
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: First group: Pyfazimine 100mg group, 12 cases. Second group: Pyfazimine 200mg group, 12 cases. Third group: Pyfazimine 300mg group, 12 cases. Forth gourp: Pyrazinamide 1500mg group, 10 cases. Fifth group: Pyfazimine 200mg + Pyrazinamide 1500mg group, 10 cases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First group (Experimental): Pyfazimine 100mg group, 12 cases.
  Interventions: Drug: Pyrifazimine (TBI-166)
- Second group (Experimental): Pyfazimine 200mg group, 12 cases.
  Interventions: Drug: Pyrifazimine (TBI-166)
- Third group (Experimental): Pyfazimine 300mg group, 12 cases.
  Interventions: Drug: Pyrifazimine (TBI-166)
- Forth group (Active Comparator): Pyrazinamide 1500mg group, 10 cases.
  Interventions: Drug: Pyrifazimine (TBI-166)
- Fifth group (Active Comparator): Pyfazimine 200mg + Pyrazinamide 1500mg group, 10 cases.
  Interventions: Drug: Pyrifazimine (TBI-166)

INTERVENTIONS:
Drug: Pyrifazimine (TBI-166) — The new drug pyrifazimine (previous name: TBI-166) is obtained by retaining the key skeleton of the lead drug clofazimine which can exert its efficacy and modification by introducing moderate polar groups structural. While the drug has strong activity against tuberculosis-sensitive bacteria and drug-resistant bacteria in vivo and in vitro, its pharmacokinetic properties and skin staining side effects have been significantly improved compared with the lead drugs, so that the drug can achieve the goal that reducing fat solubility, accelerating metabolism in the body, reducing skin staining and reducing side effects.
  In November 2016, the new anti-drug-resistant tuberculosis drug pyrifazimine and its tablets obtained the drug clinical approval issued by the CFDA, and were approved the clinical stage research that development of drug-resistant tuberculosis adaptation.

SUMMARY:
The new drug pyrifazimine (previous name: TBI-166) developed by the Institute of Materia Medica of the Chinese Academy of Medical Sciences which is Beijing Union Pharmaceutical Second Factory relied on is obtained by retaining the key skeleton of the lead drug clofazimine which can exert its efficacy and modification by introducing moderate polar groups structural. While the drug has strong activity against tuberculosis-sensitive bacteria and drug-resistant bacteria in vivo and in vitro, its pharmacokinetic properties and skin staining side effects have been significantly improved compared with the lead drugs, so that the drug can achieve the goal that reducing fat solubility, accelerating metabolism in the body, reducing skin staining and reducing side effects. In addition, pyrifazimine has a weak effect on liver drug enzymes, and is suitable for combined use in the clinical treatment of tuberculosis. The development of the drug is expected to provide a new method for the clinical treatment of drug-resistant tuberculosis, benefit patients, and produce good social benefits.

In November 2016, the new anti-drug-resistant tuberculosis drug pyrifazimine and its tablets (formerly chemical drug registration classification 1.1) obtained the drug clinical approval issued by the CFDA (batch number: 2016L10025/2016L09987), and were approved the clinical stage research that development of drug-resistant tuberculosis adaptation.

In accordance with relevant requirements of drug registration regulations, technical guidelines, etc., this project has completed the safety, tolerability, and pharmacokinetic clinical trials of a single dose of pyrifazimine tablets in healthy subjects, i.e. Phase Ia clinical trials test.

ELIGIBILITY:
Inclusion Criteria:

* (Those who must meet all the selection criteria can enter the group)

  1. People who volunteer to participate in this trial and sign an informed consent form;
  2. The range of the age is from 18 to 65 years old, regardless of gender;
  3. The weight range of the patient who wear lightweight clothing and no shoes is from 40 to 90 Kg;
  4. The patient is diagnosed with (initial treatment) tuberculosis, and the untreated sputum smear is 2+ or 2 times 1+ or more;
  5. Chest x-ray examination results are consistent with tuberculosis;
  6. Molecular tests show positive for Mycobacterium tuberculosis (e.g. GeneXpert or Hain) or positive for sputum culture;
  7. Women in the reproductive period have a negative urine pregnancy test and agree to use high-efficiency contraception during the study period;
  8. Male patients must agree to use appropriate contraceptive methods.

Exclusion Criteria:

* (Meet any of the following criteria will be excluded)

  1. Those who cannot tolerate treatment delay;
  2. Those who have used any drugs that are effective against Mycobacterium tuberculosis within 3 months before screening;
  3. History of allergy to clofazimine, rifamycin and its derivatives, isoniazid, pyrazinamide or ethambutol;
  4. Use any drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes within 30 days before administration (Including but not limited to quinidine, tyramine, ketoconazole, fluconazole, testosterone, quinine, progesterone, Methitione, phenpromazine, doxorubicin, trilithomycin, erythromycin, cocaine, furanilide, cimetidine, dextromethorphan);
  5. Resistance to isoniazid and rifampicin;
  6. Any disease or symptom that contradicts the use of rifampicin, isoniazid, pyrazinamide or ethambutol;
  7. Severe extrapulmonary tuberculosis (blood disseminated tuberculosis, digestive system tuberculosis, genitourinary tuberculosis, bone and joint tuberculosis, tuberculosis meningitis, etc.);
  8. There is evidence of silicosis, pulmonary fibrosis or other lung diseases considered by researchers to be serious (except tuberculosis);
  9. The patient has chronic obstructive pulmonary disease or asthma;
  10. Any clinically relevant concomitant circumstances or renal impairment characterized by serum creatinine level ≥1.5xULN, or liver damage with ALT and/or AST level ≥3×ULN and/or GGT level ≥3×ULN within the laboratory reference range;
  11. History of alcohol abuse [weekly alcohol intake is greater than 21 units/week (male) and 14 units/week (female) (1 unit=360mL beer; or 150mL glucose wine; or 45mL white wine)], or the subject is unwilling to stop drinking from 24 hours before the start of the study to the end of the study, or had a positive alcohol breath test at the time of enrollment;
  12. Subjects with liver, kidney, metabolism, autoimmune diseases, neurological, mental, blood system diseases, malignant tumors, long-term immunosuppressive agents;
  13. People with a history of drug abuse or a positive urine drug screening;
  14. Screening positive for hepatitis B, HIV, HCV virus and Treponema pallidum antibody;
  15. Those who have a history of fainting needles and are judged to be clinically significant by the investigator;
  16. Participated in clinical research of other drugs or devices three months before the start of the trial;
  17. The subject has the following characteristics at the time of screening (according to the measurement and reading of the central electrocardiogram):

  <!-- -->

  1. The QT/QTc interval is significantly prolonged, for example, the QTcF (Fridericia correction) or QTcB (Bazett correction) interval is confirmed to be >450 ms during screening;
  2. Has a history of Ventricular tachycardia torsades de pointes, such as heart failure, hypokalemia, long QT syndrome, etc.;
  3. Uses any drug known to extend the QTc interval 30 doses before the medication. (Not limited to amiodarone, bepridil, chloroquine, chlorpromazine, cisapride, cyclobenzaprine, clarithromycin, dipyrazine, doperidol, erythromycin, fluorine alcohol, Haloperidol, ibutilide, levamisole, methadone, mesalamide, pimozine, procaine, quinine, sotalol, sparfloxacin, thiazide);
  4. The investigator judges that any ECG abnormalities of clinical significance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
EBA | The change of TB bacterium burden in sputum from Day 0 to Day 7 and/or Day 14
  Early bactericidal activity (EBA), counted by daily log (CFU) change

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Zhengzhou Sixth People's Hospital, Zhengzhou, Henan
  - Shandong Chest Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No